CLINICAL TRIAL: NCT06380608
Title: Assessing Levels of Fear and Anxiety and Monitoring Wound Healing Among Patients Who Are About to Undergo Wisdom Tooth Extraction Surgery or Jaw Implant Surgery Under Local Anesthesia Versus General Anesthesia
Brief Title: Levels of Fear, Anxiety and Wound Healing Among Aental Surgery Patients Under Local Versus General Anesthesia
Status: Recruiting | Type: Observational
Sponsor: Zoya Haitov Ben Zikri (Other Government)
Responsible Party: Sponsor-Investigator, Zoya Haitov Ben Zikri, Director of the anesthesia department, Assaf-Harofeh Medical Center
Organization: Assaf-Harofeh Medical Center (Other Government)
Other Study IDs: 0047-23-ASF
Record Dates: First submitted 2023-09-07; First posted 2024-04-24 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Wisdom Teeth Extraction or Jaw Implant
MeSH Terms: interventions — Anesthesia, Local; Anesthesia, General

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Weeks
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Local Anesthesia: Patients who will undergo a dental surgery under local anesthesia
  Interventions: Procedure: Local anesthesia
- General anesthesia: Patients who will undergo a dental surgery under general anesthesia
  Interventions: Procedure: General anesthesia

INTERVENTIONS:
Procedure: Local anesthesia — Patients who will undergo a dental surgery under local anesthesia
  Groups: Local Anesthesia
Procedure: General anesthesia — Patients who will undergo a dental surgery under general anesthesia
  Groups: General anesthesia

SUMMARY:
Tooth extraction is one of the most common procedures in dentistry. Surgical extraction of damaged wisdom teeth involves bone resection and injury to the soft tissue. Dental care often evokes high levels of anxiety.In addition, stress causes poor regulation of endocrine, autocrine and paracrine systems during the three stages of wound healing of the soft oral tissues. Therefore, special considerations are necessary when performing dental surgery on highly stressed patients. One of the options used in the last decade is to perform this procedure under general anesthesia.

A stress response stimulates the secretion of cortisol hormone. Cortisol levels were found to be significantly higher before dental surgery, while after the operation the hormone level dropped significantly.

The aim of the study is to assess the level of anxiety/fear and monitor the wound healing process among patients who are about to undergo surgery to remove wisdom teeth or no more than 3 jaw implants under local anesthesia in the dental clinic compared to patients who are about to undergo the same surgery under general anesthesia.

DETAILED DESCRIPTION:
The study will include subjects who are about to undergo extraction of wisdom teeth or no more than 3 implants in the jaw under local anesthesia in the dental clinic or under general anesthesia in a hospital operating room.

Patients will sign an informed consent form before entering the study. The various measurements of the study will include -

* Level of free cortisol in saliva. Saliva collection will be performed between 9 am and 12 noon. 2 ml of saliva will be collected from the patient by asking the patient to spit into a disposable container.
* The level of fear of pain - will be measured using the Fear of Pain Questionnaire- (FPQ-III), which is widely used to assess the fear of pain. This questionnaire contains 30 items.
* The level of fear of dental pain - in this study the short version of the fear of dental pain questionnaire - FDPQ will be used to assess the fear of pain related to a variety of dental procedures.
* Level of dental anxiety - dental anxiety will be assessed by the dental anxiety scale of The DAS Corah consisting of four questions about different dental conditions
* To monitor the inflammation, the inflammatory proliferation scale (IPR) will be used to monitor the wound healing process.

The study includes 5 visits:

Visit 1: 5-7 days before surgery - in the waiting room of the dental clinic

* Patients will sign an informed consent form.
* The patients will answer a questionnaire regarding their demographic characteristics (age, sex, marital status, income, education, medical and dental history).
* The patients will fill out a fear of pain questionnaire, a fear of toothache questionnaire and a fear of dental care questionnaire
* The dentist will answer a questionnaire about the dental and medical history of the patients, the condition of the teeth, the type of anesthesia and the type of treatment that will be performed under anesthesia.
* A saliva sample will be collected from the patients between 9:00 and 12:00 for cortisol level measurements.

Visit 2: On the day of surgery, in the waiting room of the dental clinic or the operating room (depending on the type of anesthesia planned) before the procedure-

* The patients will fill out a fear of pain questionnaire, a fear of dental pain questionnaire and a dental anxiety anxiety questionnaire.
* A saliva sample will be collected from the patients between 9:00 and 12:00 for cortisol level measurements.

Visit 3: 5 days after the operation - in the waiting room of the dental clinic

* The patients will fill out a fear of pain questionnaire, a fear of toothache questionnaire and a fear of dental care questionnaire.
* The dentist about the complications and claims reported by the patient
* A saliva sample will be collected from the patients between 9:00 and 12:00 for cortisol level measurements.
* The surgeon will complete the IPR. Visit 4: 14 days after surgery
* The surgeon will complete the IPR. Visit 5: 6 weeks after surgery
* The surgeon will complete the IPR.

ELIGIBILITY:
Inclusion Criteria:

* Age - from ≥ 18 years,

  * ASA 1- or 2,
  * Signing a written informed consent before starting all procedures related to the research,
  * Ability to cooperate with the researcher and meet the research requirements.

Exclusion Criteria:

* Not relevant

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who are about to undergo a dental surgery under local or general anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 46 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Fear and anxiety | 7-8 weeks
  The level of fear of pain will be measured using the Fear of Pain Questionnaire This questionnaire contains 30 items. Each question presents a pain-related situation, and participants are asked to rate FOP on a 5-point Likert scale (not afraid at all, 5= extremely afraid) The level of fear of dental pain will be measured by the short version of the fear of dental pain questionnaire - FDPQ. The questionnaire consists of 18 items and assesses fear of pain associated with a variety of dental procedures. Each item is answered on a rating of 1 (no fear) to 5 (extreme fear), resulting in a possible total score of 18-90.
  Dental anxiety level - dental anxiety will be assessed by the dental anxiety scale of The DAS Corah. The questionnaire consists of 4 items describing successively situations related to dental treatment: For each item, the subject has to respond using a five point scale.
Wound heeling | 7-8 weeks
  The Inflammatory Proliferative Remodeling (IPR) Wound Healing Scale will be used in order to evaluate the wound healing. The scale is divided into three subscales corresponding to the three phases of wound healing: The inflammatory phase (days 3-5 postoperatively), The proliferative phase (14 days postoperatively) and the remodeling phase (6 weeks postoperatively). Each clinical manifestation was scored 0 or 1, yielding three subscale scores ranging from 0-8, 0-5, and 0-3, accordingly.

CONTACTS AND LOCATIONS:
Overall Officials: Zoia Haitov Ben Zikri, MD, Principal Investigator — Assaf-Harofeh Medical Center
Locations (1):
- Shamir (Asaf Harofe) Medical center, Be’er Ya‘aqov, Israel

IPD SHARING:
Plan to Share IPD: No